CLINICAL TRIAL: NCT01555385
Title: The Effects of Nutritive and Non-nutritive Breakfast on Subjective Mental Workload During Multitasking - a Pilot Study in Healthy Volunteers
Brief Title: The Effects of Breakfast on Mental Workload
Acronym: AivoPro1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Finnish Institute of Occupational Health (Other); SalWe Ltd. (Industry)
Responsible Party: Principal Investigator, Katri Peuhkuri, Principal investigator, postdoctoral reseacher, authorized nutritionist, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UH-SHOK-001
Record Dates: First submitted 2012-03-14; First posted 2012-03-15 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Subjects
Keywords: Mental workload; Multitasking; Protein; Tryptophan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dietary supplement: high-protein breakfast (Active Comparator): high-protein juice
  Interventions: Dietary Supplement: Breakfast juice
- Dietary supplement: high-carbohydrate breakfast (Active Comparator): high-carbohydrate juice
  Interventions: Dietary Supplement: Breakfast juice
- Dietary supplement: low energy breakfast (Placebo Comparator): low-calorie juice
  Interventions: Dietary Supplement: Breakfast juice

INTERVENTIONS:
Dietary Supplement: Breakfast juice — single dose (300 ml) in the morning of study day, 3 separate sessions (high-protein vs. high-carbohydrate vs. low-calorie juice), total duration 3 weeks

SUMMARY:
The aim of the study is to investigate the influence of nutritive (high-protein or high-carbohydrate) and non-nutritive (low energy) breakfast on psychological and physiological responses of mental workload during multitasking in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* eats usually breakfast
* use computer mouse with right hand
* normal sleep-wake rhythm between 9 pm and 8 am
* in females hormonal contraception

Exclusion Criteria:

* gastrointestinal disease, diabetes or any other significant major medical morbidity
* milk allergy
* lactose intolerance
* smoking
* excess use of alcohol, coffee, tea, cola drinks (> 10 doses/day)
* pregnancy and breast feeding
* no medication or dietary supplements influencing measured responses
* BMI > 30 kg/m2 or < 18 kg/m2

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Brain measures of mental workload (ERP 300 amplitude and latency) and heart rate | 1 day

SECONDARY OUTCOMES:
Subjective mental workload and mood measurement assessed using visual analogue scale in response to test meal. | 1 day
cognitive function measurements | 1 day
Blood concentration of glucose | 1 day
salivary cortisol | 1 day
Blood concentration of tryptophan in relation to other large neutral amino acids | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- University of Helsinki, Institute of Biomedicine, Helsinki, Finland